CLINICAL TRIAL: NCT05341778
Title: Effects of Pilates Exercises Versus Pelvic Floor Muscle Exercises Among Elderly Women With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Collaborators: The Institute of Physical Medicine and Rehabilitation (Other)
Responsible Party: Principal Investigator, Humera Ahmed, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAhmed
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Urinary Incontinence
Keywords: Urinary incontinence; Older females; Pelvic floor disorders; Urination; Quality of life
MeSH Terms: conditions — Urinary Incontinence; Pelvic Floor Disorders | interventions — Surgical Instruments

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the type of treatment provided to the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercises (Experimental): The Pilates method's exercises emphasize breathing and the activation of the deep stabilizing muscles of the trunk in coordination with the PFM. The pilates method consists of exercises that emphasize pelvic stability, mobility, and body alignment. PMFE are performed in tandem with breathing, with concurrent trunk muscle recruitment in various positions.
  Interventions: Other: Shoulder bridge; Other: Clam shell; Other: Scissors; Other: Adductor squeeze; Other: Pelvic clock supine; Device: Electrical muscle stimulation
- Pelvic floor exercise (Active Comparator): These exercises are intended to strengthen weak perineal and pelvic floor muscles.
  Interventions: Other: Clam shell; Other: Adductor squeeze; Other: urine hold and tummy tuck in; Other: Bridging; Other: Split table top; Device: Electrical muscle stimulation

INTERVENTIONS:
Other: Shoulder bridge — The shoulder bridge is great for, strengthening your gluteal muscles, quadriceps, hamstrings, pelvic floor, abdominals and back muscles; most notably the tiny ones which control movement of each individual vertebrae and can weaken after episodes of back pain.
  Arms: Pilates exercises
Other: Clam shell — Scissors is an abdominal exercise that strengthens the transverse abdominals, helping flatten your belly and strengthen your entire core. Scissors is not only a core strength move, but it is also a great stretch for your hamstrings and your lower back.
Other: Scissors — Scissors is an abdominal exercise that strengthens the transverse abdominals, helping flatten your belly and strengthen your entire core. Scissors is not only a core strength move, but it is also a great stretch for your hamstrings and your lower back.
  Arms: Pilates exercises
Other: Adductor squeeze — Adductor Squeeze exercise The SQ exercise is an isometric hip adduction exercise with the player holding a ball between their knees.
Other: Pelvic clock supine — The pelvic clock is a brilliant exercise to help achieve flexibility and strength in the lower back, pelvic floor, and core-in order to prevent pain and injury.
  Arms: Pilates exercises
Other: urine hold and tummy tuck in — During tummy tuck patients are able to strategically tighten and reinforce the muscles around the pelvic floor, urethra, and other structures. This increased strength and support greatly reduces stress urinary incontinence
  Arms: Pelvic floor exercise
Other: Bridging — A bridge exercise isolates and strengthens your gluteus (butt) muscles - the gluteus maximus, medius and minimus - and hamstrings, which are the main muscles that make up the posterior chain. It is done by lying on your back with your knees bent, feet flat on the ground and at a comfortable distance from your butt.
  Arms: Pelvic floor exercise
Other: Split table top — To strengthen your abs, shoulders, arms and legs. The most important part of this move is to contract your abs fully before you start to lower your hips
  Arms: Pelvic floor exercise
Device: Electrical muscle stimulation — Electric stimulation works by mimicking the natural way by which the body exercises its muscles. The electrodes attached to the skin deliver impulses that make the muscles contract. It is beneficial in increasing the patient's range of motion and improves the circulation of the body.

SUMMARY:
To compare the effects of Pilates exercises versus pelvic floor muscle exercises among elderly women with urinary incontinence. The study is a single-blinded randomized clinical trial. 70 patients(calculated through PASS version 15 software) will be selected. Subjects will be screened whether they met inclusion and exclusion criteria. The participants for this study will be elderly women with urinary incontinence. The participants will be recruited from SIPMR and Civil hospital Karachi. The initial assessment will be done by Medical Consultant. Patients must fulfill inclusion criteria. Consent must be taken from each patient and samples will be collected in the given time frame and patients will be randomly assigned(through a randomization sheet) to the treatment groups. Treatment group 1 will be doing Pilates exercises and treatment group 2 will be doing Pelvic floor muscle exercises. EMS will be given to both treatment groups. A voiding diary, Stamey's urinary incontinence system, and IQOL questionnaire will be used at baseline assessment and at the end of treatment sessions. 12 treatment sessions will be given, 3 visits each week for 4 weeks. The data will be analyzed on SPSS version 21. : Non-probability purposive sampling technique will be used for selecting individuals. Percentages and frequencies will be calculated for categorical variables and parametric and nonparametric tests will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Elderly females from an outpatient setting of Sindh Institute of physical medicine and rehabilitation and civil hospital Karachi.
* Patients aged ≥60 years.
* Experienced stress or mixed urinary incontinence symptoms at least 3 times/ week for 3 months or more.

Exclusion Criteria:

* Have limited mobility (unable to move without crutches, walker, or a cane).
* Have untreated chronic constipation or have experienced any stool or mucus leakage.
* Organ prolapse surgery within the last year.
* In the last 3 months, any active urinary or vaginal infection.
* Malignancy

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility will be based on self-representation of gender identity.
Enrollment: 70 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Change in volume of urine in millilitre on Voiding Diary after 4 weeks | baseline and after 4 weeks
  It will be recorded by patient in millilitre in a marked beaker. Increase in millilitre suggests increase in volume of urine.
Change in intensity and frequency of urine leakage on Voiding Diary after 4 weeks | baseline and after 4 weeks
  It will be recorded by patient with yes or no option. Increase in ticks on yes options suggests increase in intensity and frequency of urine leakage.
Change in the number of pads on Voiding Diary after 4 weeks. | baseline and after 4 weeks
  It will be recorded by patient with the symbol P if yes and blank if No. Increase in written symbol P suggests increased number of pads.
Change in frequency and grading of urgency on Voiding Diary after 4 weeks | baseline and after 4 weeks
  It will be recorded by patient with grades 0=little, +=mild, ++=extreme urgency. The more the score the worst the urinary incontinence is.
Change in urine incontinence on Stamey's incontinence scoring system after 4 weeks | baseline and after 4 weeks
  It is based on the patient's incontinence history alone. It will be graded from 0=no incontinence to 3=total incontinece at all times.The higher the score the more severity of urinary incontinence is

SECONDARY OUTCOMES:
Change in Quality of life on Quality of life measures questionnaire scores after 4 weeks | baseline and after 4 week
  All the participants will complete an incontinence-related quality of life questionnaire to assess the quality of life of patients suffering from urinary incontinence.Higher the scores, the higher will be quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Aftab Ahmed Mirza Baig, MSAPT, Study Director — Sindh Institute of Physical Medicine and Rehabilitation; Humera Ahmed, DPT, Principal Investigator — Dow University of Health Sciences; Rabail Rani Soomro, MSPT, Study Director — Sindh Institute of Physical Medicine and Rehabilitation
Locations (1):
- Humera Ahmed, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD yet.